CLINICAL TRIAL: NCT06891924
Title: Clinical Study on Pre-operative Intervention With Products to Mitigate Skin Discomfort During Aesthetic Medicine
Brief Title: A Clinical Study on Pre-operative Intervention With Products During Aesthetic Medicine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Botanee Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Botanee-252003
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Skin Aging; Skin Condition; Skin Manifestations
MeSH Terms: conditions — Skin Diseases; Skin Manifestations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formulation containing MLYAAT-1002® Composition (Active Comparator): Before the Fotana4D Pro® treatment, daily use of the formulation containing MLYAAT-1002® for 14 days: apply one pump of the formulation to the test side of the face twice daily.
  Interventions: Combination Product: 14-day daily pre-operative application of the formulations containing MLYAAT-1002® before Fotona4D treatment
- Blank formulation without MLYAAT-1002® Composition (Placebo Comparator): Before the Fotana4D Pro® treatment, daily use of the formulation without MLYAAT-1002® for 14 days: apply one pump of the formulation to the control side of the face twice daily.
  Interventions: Combination Product: 14-day daily pre-operative application of the formulations without MLYAAT-1002® before Fotona4D treatment

INTERVENTIONS:
Combination Product: 14-day daily pre-operative application of the formulations containing MLYAAT-1002® before Fotona4D treatment — All enrolled subjects will complete a 14-day washout period followed by a 14-day run-in phase prior to Fotona 4D® laser treatment. During the initial washout phase, participants will exclusively use basic skincare products: sunscreen, cleansing foam, and moisturizing emulsion. Then the subjects will apply the formulations containing MLYAAT-1002® of the active comparator to randomly assigned split-face (the treatment side) for the subsequent 14-day period. Following completion of the product application regimen, all participants will undergo a single session of Fotona 4D laser therapy.
  Arms: Formulation containing MLYAAT-1002® Composition
Combination Product: 14-day daily pre-operative application of the formulations without MLYAAT-1002® before Fotona4D treatment — All enrolled subjects will complete a 14-day washout period followed by a 14-day run-in phase prior to Fotona 4D® laser treatment. During the initial washout phase, participants will exclusively use basic skincare products: sunscreen, cleansing foam, and moisturizing emulsion. Then the subjects will apply the formulations without MLYAAT-1002® of the placebo comparator to randomly assigned split-face (the control side) for the subsequent 14-day period. Following completion of the product application regimen, all participants will undergo a single session of Fotona 4D laser therapy.
  Arms: Blank formulation without MLYAAT-1002® Composition

SUMMARY:
This clinical trial aims to evaluate whether a 14-day pre-operative application of the test product (containing MLYAAT-1002®, a proprietary anti-aging complex) can mitigate skin discomfort during Fotona 4D laser therapy (Frac3 and Piano modes) by comparing clinical evaluation, skin attributes measurement and subject self-assessment.

ELIGIBILITY:
Inclusion Criteria:

* health females aged 35-60;
* subjects with rough dark, loose fine lines;
* no history of cosmetic allergies;
* subjects are willing to use the test serum on split-face for 28 days;
* subjects are willing to suffer the Fotona 4D treatment (Frac3 and Piano modes) on the face;
* subjects are willing to use the basic skincare products for 28 days, and acceptable for split-face use of the test products or the control product for 14 days;
* written informed consent and portrait right consent were obtained from all participants before study entry.

Exclusion Criteria:

* anyone who is pregnant, nursing an infant, or planning a pregnancy during the study;
* subjects with known allergies or sensitivities to the ingredients in any of the study products;
* any symptoms of facial flushing, erythema, papules, desquamation, or edema as evaluated by a physician prior to initial screening or Fotona4D Pro treatment;
* unhealed skin lesions;
* participated in any other clinical trial within one month;
* received facial skin treatments including but not limited to lasers, chemical peels, and dermal fillers within one month;
* taken/injected anti-allergy medication in the past one month;
* participants in other clinical trials at the same time;
* any subjects that the investigator considers ineligible.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
changes in the percentage of area in the red zone of facial skin | Baseline (before Fotona 4D treatment), T30min (30 minutes after Fotona 4D treatment), T2h (2 hours after Fotona 4D treatment)
  capturing facial images by VISIA-CR (CANFIELD, America) and analysis the percentage of area in the red zone.
Self-assessment of the facial state questionnaire | Baseline (before Fotona 4D treatment), Timm (immediately after Fotona 4D treatment), T30min (30 minutes after Fotona 4D treatment), T2h (2 hours after Fotona 4D treatment)
  Subjects rated the burning sensation, picotement, pruritus, dysesthesia, tightness,on a five-point scale: 0=Asymptomatic;1=Very mild;2=mild;3=moderate;4=severe

SECONDARY OUTCOMES:
changes in transepidermal water loss (TEWL) of facial skin | D-14(14 days before Fotona 4D treatment), Baseline (before Fotona 4D treatment), T30min (30 minutes after Fotona 4D treatment), T2h (2 hours after Fotona 4D treatment)
  measuring the loss of water that passes from inside a body through the epidermis to the surrounding atmosphere by Vapometer.
changes in skin stratum corneum water content | D-14(14 days before Fotona 4D treatment), Baseline (before Fotona 4D treatment), T30min (30 minutes after Fotona 4D treatment), T2h (2 hours after Fotona 4D treatment)
  measuring skin stratum corneum water content by Corneometer CM825 (Courage&Khazaka，Germany).

IPD SHARING:
Plan to Share IPD: No